CLINICAL TRIAL: NCT01390246
Title: Bupropion for Smoking Cessation During Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-217; R01DA030998 (NIH)
Record Dates: First submitted 2011-06-08; First posted 2011-07-08 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2018-02

CONDITIONS: Pregnancy Related; Tobacco Use Disorder
Keywords: Pregnancy; Tobacco use disorder; Smoking cessation; Bupropion SR; Zyban
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Bupropion; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion SR + cessation counseling (Active Comparator): Bupropion SR and smoking cessation counseling Subjects received Bupropion SR 150 mg tablet orally twice daily (BID) for 12 weeks. Subjects were instructed to begin using study medication (bupropion SR 150 mg orally for 3 days, then BID for 4 days) on study visit day 1, which was approximately 1 week prior to their quit date. Thereafter, they were continued to dose Bupropion SR 150 mg tablet orally BID for a total medication treatment of 12 full weeks.
  Smoking cessation counseling included 35-minute counseling sessions at each of the first 2 visits and 10 minutes of smoking cessation counseling at subsequent visits, provided by the trained study nurse.
  Interventions: Drug: Bupropion SR; Behavioral: Smoking Cessation Counseling
- Placebo + cessation counseling (Placebo Comparator): Placebo and smoking cessation counseling Subjects received matching Bupropion SR placebo tablet orally twice daily (BID) for 12 weeks. Subjects were instructed to begin using study medication (matched placebo tablets orally for 3 days, then BID for 4 days) on study visit day 1, which was approximately 1 week prior to their quit date. Thereafter, they were continued to dose matching Bupropion SR placebo tablet orally BID for a total medication treatment of 12 full weeks of therapy.
  Smoking cessation counseling included 35-minute counseling sessions at each of the first 2 visits and 10 minutes of smoking cessation counseling at subsequent visits, provided by the trained study nurse.
  Interventions: Behavioral: Smoking Cessation Counseling; Drug: Placebo

INTERVENTIONS:
Drug: Bupropion SR — Bupropion SR 150 mg tablet
  Other Names: Zyban; buproban
  Arms: Bupropion SR + cessation counseling
Behavioral: Smoking Cessation Counseling — 35-min counseling by trained research nurse
  Other Names: Behavioral counseling
Drug: Placebo — Matching Bupropion SR placebo tablet
  Other Names: Control
  Arms: Placebo + cessation counseling

SUMMARY:
This is a prospective, double-blind placebo-controlled randomized pilot trial of the preliminary safety and efficacy of bupropion SR in combination with behavioral counseling for smoking cessation during pregnancy.

DETAILED DESCRIPTION:
This is a prospective, double-blind placebo-controlled randomized pilot trial of the preliminary safety and efficacy of bupropion SR in combination with behavioral counseling for smoking cessation during pregnancy. A total of 150 pregnant smokers will receive medication (75) or placebo (75) for 12 weeks. Compassionate care/continuance of therapy will be available to pregnant subjects. Women who relapse to smoking postpartum will be offered an additional course of medication treatment. All subjects regardless of adherence with 12 week study drug administration period and smoking habits during pregnancy will be followed through the duration of their pregnancy, delivery, and 6-month postpartum period. Subject participation will begin between 13-30 wks of gestation and end 6 months postpartum. Participation will be ten (10) to thirteen(13) months in length.

ELIGIBILITY:
Inclusion Criteria:

* smoking at least 10 CPD prior to pregnancy and 5 CPD for the preceding 7 days
* 13-30 weeks gestation
* ≥18 years of age
* able to speak English or Spanish
* intent to carry pregnancy to term
* stable residence

Exclusion Criteria:

* current illicit drug or alcohol abuse or dependence
* twins or other multiple gestation
* treatment for psychiatric disorder within the last 6 months
* unstable medical problems (eg, hypertension (BP>140/90), preeclampsia, threatened abortion, hyperemesis gravidarum)
* known congenital abnormality
* seizure disorder
* use of psychotropic medication
* use of medication known to lower the seizure threshold
* anorexia/bulimia
* a personal history of closed head trauma with > 30 minutes of loss of consciousness or amnesia or resulting in skull fracture or subdural hematoma/brain contusion
* use of any other smoking cessation treatment in the past 30 days
* current enrollment in methadone treatment program
* prior pregnancy with preeclampsia diagnosis
* chronic hypertension (past history or current diagnosis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary DV Hankins, MD, Principal Investigator — The University of Texas Medical Branch, Galveston; Tatiana Nanovskaya, PhD, Principal Investigator — The University of Texas Medical Branch, Galveston; Cheryl Onken, MD, MPH, Principal Investigator — UConn Health; Mahmoud Ahmed, PhD, Principal Investigator — The University of Texas Medical Branch, Galveston; Shannon Clark, MD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch at Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Result] Nanovskaya TN, Oncken C, Fokina VM, Feinn RS, Clark SM, West H, Jain SK, Ahmed MS, Hankins GDV. Bupropion sustained release for pregnant smokers: a randomized, placebo-controlled trial. Am J Obstet Gynecol. 2017 Apr;216(4):420.e1-420.e9. doi: 10.1016/j.ajog.2016.11.1036. Epub 2016 Nov 25. PMID 27890648

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant smokers were recruited through the UTMB Ob/Gyn Department clinics and Regional Maternal Child Health Program (RMCHP) clinics. The study was also advertised through printed flyers, posters, and electronic media in clinic waiting areas. UTMB OB providers were notified of the study as well to refer potential participants.
Pre-assignment Details: Psychological screening using the PRIME MD survey was administered after enrollment at the first Study Visit. Using the score, subjects with evidence of major depression or any other severe, acute psychiatric symptom (eg, psychosis) were considered screen failures and referred back to their prenatal provider for treatment.
Groups:
- Bupropion SR: Subjects received 150 mg tablet bupropion SR orally once daily for three days followed by twice daily for a total medication treatment of 12 weeks.
  Subjects also received behavioral interventions, which included 35-minute counseling sessions at each of the first 2 visits (enrollment and on the quit day) and 10 minutes of smoking cessation counseling at subsequent visits.
- Placebo: Subjects received matched bupropion SR placebo tablet orally once daily for three days followed by twice daily for a total medication treatment of 12 weeks.
  Subjects also received behavioral interventions, which included 35-minute counseling sessions at each of the first 2 visits (enrollment and on the quit day) and 10 minutes of smoking cessation counseling at subsequent visits.
Period: Overall Study
Arm/Group | Bupropion SR | Placebo
Started | 30 | 35
Visit 2: Quit Day | 24 | 24
Visit 6: End of Treatment | 15 | 15
Visit 7: 36-38 Weeks Gestation | 10 | 10
Completed | 10 | 10
Not Completed | 20 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion SR | Placebo | Total
Number analyzed (Participants) | 30 | 35 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 35 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (5.56) | 27.5 (6.52) | 26.2 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 65
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 25 | 30 | 55
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 13 | 16
  White | 27 | 22 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 35 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in Cigarette Craving and Total Nicotine Withdrawal Symptoms Between Groups During Medication Treatment
Description: Cigarette craving and withdrawal symptoms were assessed by the Minnesota Nicotine Withdrawal Scale (MNWS). MNWS consists of 7 objectives (e.g., irritability, anxious, depressed mood, difficulty concentrating, increased appetite, insomnia, restless). Subjects were given a score on each item on a scale of 0 (not present) to 4 (severe). Summed (total) score excluding craving represent subject's symptoms of tobacco withdrawal, ranging from 0 to 28. We calculated a craving for tobacco score and a total score of withdrawal symptoms excluding craving. The higher score represent more sever craving and withdrawal.
Time Frame: During treatment: Visits 2-6 (time period between 2nd and 12th week of therapy)
Measure: Mean (Standard Deviation); unit: MNWS Score
Arm/Group | Bupropion SR | Placebo
Number analyzed (Participants) | 24 | 24
MNWS Score
  Craving for tobacco | 1.50 (1.11) | 2.07 (1.23)
  Total score of withdrawal excluding craving | 3.77 (4.27) | 5.35 (5.14)

2. Primary Outcome: Change in Cigarette Craving and Total Nicotine Withdrawal Symptoms Between Groups on the Quit Date
Description: as for outcome 1
Time Frame: Quit date, visit 2 (one week after starting the 12-week course of therapy)
Measure: Mean (Standard Deviation); unit: MNWS Score
Arm/Group | Bupropion SR | Placebo
Number analyzed (Participants) | 24 | 24
MNWS Score
  Craving for tobacco | 2.04 (1.08) | 2.33 (1.31)
  Total score of withdrawal excluding craving | 4.75 (4.87) | 4.88 (4.61)

3. Primary Outcome: Number of Participants With 7-day Point Prevalence Smoking Abstinence at the End of Medication Treatment (Visit 6)
Description: The accuracy of self-reported smoking abstinence during study visits was confirmed by an exhaled carbon monoxide (CO) levels and by urinary cotinine levels. 7-day point prevalence abstinence was defined as no cigarettes (not even a puff) in the last 7 days, levels of (CO) in exhaled air < 4 ppm, and concentrations of cotinine in urine < 50 ng/mL. At every visit, a research nurse monitored the smoking status of all subjects (amount of cigarettes per day, exhaled CO). Exhaled CO was measured using a Vitalograph carbon monoxide monitor (Lenexa, KS) according to the manufacturer's recommendations. A urine sample was collected at each visit and cotinine in urine was quantified using the validated liquid chromatography-mass spectrometry (LC/MS) method. We calculated the total number of abstinent subjects. The higher the number the better outcome.
Time Frame: Visit 6 (end of 12 weeks of medication therapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion SR | Placebo
Number analyzed (Participants) | 30 | 35
Participants | 5 | 1

4. Primary Outcome: Number of Participants With 7-day Point Prevalence Smoking Abstinence at the End of Pregnancy (Visit 7)
Description: as for outcome 3
Time Frame: End of pregnancy (visit 7) is a time period between 36.0-38.6 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion SR | Placebo
Number analyzed (Participants) | 30 | 35
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: For each pregnant woman, adverse events were assessed from enrollment through completion (or six months post partum). Neonatal adverse events were assessed at delivery and through infant discharge.
Description: We monitored for maternal AEs that could be related to bupropion, such as seizures, consistent BP >140/90 mm Hg, headache, insomnia, rhinitis, dry mouth, and anxiety. We defined a priori which AEs would be considered fetal and neonatal SAEs: intrauterine fetal demise, preterm delivery <34 weeks, clinically suspected fetal growth restriction, congenital malformations, cardiovascular anomalies, low birthweight (<10%), Apgar scores <7 at 5 minutes, and neonatal length of hospital stay >3 days.
Arm/Group | Bupropion SR | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/35
Serious Adverse Events (participants affected / at risk) | 2/30 | 5/35
Other Adverse Events (participants affected / at risk) | 14/30 | 8/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion SR (N=30) | Placebo (N=35)
Infant stay in NICU >3 days due to premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 4
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Cord blood pH <7.01 (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Gestational Diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion SR (N=30) | Placebo (N=35)
Headache (Nervous system disorders) | 12 | 6
Difficulty sleeping (Nervous system disorders) | 10 | 7
Rhinorhea- Runny Nose (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Dry mouth (Gastrointestinal disorders) | 13 | 7
Anxiety (Psychiatric disorders) | 14 | 6

LIMITATIONS AND CAVEATS:
Factors affecting enrollment included social stigma of prenatal smoking and use of medications; high rate of early withdrawal/lost to follow since longitudinal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No